CLINICAL TRIAL: NCT04165577
Title: Modulating Prefrontal Circuits Underlying Behavioral Flexibility in OCD: A TMS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1901-003
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Arms denoted as open-label do not include masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (7):
- OCD, Active TMS (Experimental): Participants with OCD who receive active rTMS
  Interventions: Device: rTMS
- OCD, Sham TMS (Sham Comparator): Participants with OCD who receive sham rTMS
  Interventions: Device: sham rTMS
- Healthy Control, Active TMS (Other): Healthy control participants who receive active rTMS
  Interventions: Device: rTMS
- Healthy Control, Sham TMS (Other): Healthy control participants who receive sham rTMS
  Interventions: Device: sham rTMS
- Healthy Control, Active TMS (1 session) (Other): Healthy control participants who receive 1 session of active, open-label rTMS
  Interventions: Device: rTMS
- Healthy Control, Active TMS (3 sessions) (Other): Healthy control participants who receive 3 sessions of active, open-label rTMS
  Interventions: Device: rTMS
- OCD, Active TMS (3 session) (Other): Participants with OCD who receive 3 sessions of active, open-label rTMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — 1-Hz rTMS targeting frontal pole
  Arms: Healthy Control, Active TMS; Healthy Control, Active TMS (1 session); Healthy Control, Active TMS (3 sessions); OCD, Active TMS; OCD, Active TMS (3 session)
Device: sham rTMS — sham rTMS targeting frontal pole
  Arms: Healthy Control, Sham TMS; OCD, Sham TMS

SUMMARY:
This study investigates whether slow-frequency repetitive transcranial magnetic stimulation targeting frontal pole can acutely modulate brain circuits which show abnormal functioning during behavioral flexibility in obsessive-compulsive disorder, as well as performance on a behavioral task.

ELIGIBILITY:
Inclusion Criteria: OCD group

* current primary diagnosis of obsessive-compulsive disorder and Yale-Brown Obsessive Compulsive Scale total score ≥ 16;
* 18-55 years of age;
* ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent;
* either no use of psychiatric medication or stable psychiatric medication use for 6 weeks prior to study entry, limited to use of serotonin reuptake inhibitors and PRN use of benzodiazepines (other psychiatric medication use excluded), and
* right-handed.

Inclusion Criteria: Healthy Control group

* 18-55 years of age;
* ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent;
* right-handed.

Exclusion Criteria: OCD group

* active problematic substance use;
* lifetime psychosis or bipolar mood disorder or OCD beliefs of delusional nature;
* clinically significant hoarding symptoms;
* active suicidal or homicidal ideation;
* significant neurological disease or intracranial pathology;
* use of medications which increase risk for seizures during TMS;
* significant or unstable medical disorders or contraindication to TMS or MRI scan.

Exclusion Criteria: Healthy Control group

* current psychiatric diagnosis;
* lifetime psychosis, bipolar mood disorder, or OCD;
* active suicidal or homicidal ideation;
* significant neurological disease or intracranial pathology;
* use of psychiatric medications;
* use of medications which increase risk for seizures during TMS;
* significant or unstable medical disorders or contraindication to TMS or MRI scan.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Resting-state functional connectivity with ventral striatum | Before rTMS and approximately 1 day following open-label rTMS
  Resting-state functional connectivity with ventral striatum (assessed via fMRI)
Resting-state functional connectivity with dorsal striatum | Before rTMS and approximately 1 day following open-label rTMS
  Resting-state functional connectivity with dorsal striatum (assessed via fMRI)
Cognitive flexibility task performance | Before rTMS and approximately 1 day following open-label rTMS
  Behavioral performance on a cognitive flexibility task (% trials correct)

OTHER OUTCOMES:
Change in regional activation in orbitofrontal cortex | Before rTMS and within 30 minutes immediately following rTMS
  Change in task-based regional activation (assessed via functional magnetic resonance imaging; fMRI) in orbitofrontal cortex
Change in regional activation in dorsolateral prefrontal cortex | Before rTMS and within 30 minutes immediately following rTMS
  Change in task-based regional activation (assessed via fMRI) in dorsolateral prefrontal cortex
Change in regional activation in anterior cingulate cortex | Before rTMS and within 30 minutes immediately following rTMS
  Change in task-based regional activation (assessed via fMRI) in anterior cingulate cortex
Resting-state functional connectivity with ventral striatum | Before rTMS and within 30 minutes immediately following rTMS
  Resting-state functional connectivity with ventral striatum (assessed via fMRI)
Resting-state functional connectivity with dorsal striatum | Before rTMS and within 30 minutes immediately following rTMS
  Resting-state functional connectivity with dorsal striatum (assessed via fMRI)
Cognitive flexibility task performance | Before rTMS and within 30 minutes immediately following rTMS
  Behavioral performance on a cognitive flexibility task (% trials correct)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Garnaat, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States